CLINICAL TRIAL: NCT00026364
Title: A Phase I Study Of ZD1839 (Iressa) In Combination With Irinotecan, Leucovorin, And 5-Fluorouracil In Previously Untreated, Stage IV Colorectal Cancer
Brief Title: ZD 1839 Plus Combination Chemotherapy in Treating Patients With Locally Advanced, Locally Recurrent, or Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02425; DFCI-01142; NCI-3792; CDR0000069023 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2001-11-09; First posted 2003-06-25 (Estimated); Last update posted 2013-03-21 (Estimated); Status verified 2002-09

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Fluorouracil; Gefitinib; Irinotecan; Leucovorin

ARMS (1):
- Arm I (Experimental): Patients receive oral ZD 1839 daily. Beginning on day 15, patients receive irinotecan IV over 90 minutes, leucovorin calcium IV over 15 minutes, and fluorouracil IV weekly on weeks 1-2. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3-6 patients receive escalating doses of ZD 1839 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, 10 additional patients are accrued to receive treatment at the MTD.
  Interventions: Drug: fluorouracil; Drug: gefitinib; Drug: irinotecan hydrochloride; Drug: leucovorin calcium

INTERVENTIONS:
Drug: fluorouracil
Drug: gefitinib
Drug: irinotecan hydrochloride
Drug: leucovorin calcium

SUMMARY:
Phase I trial to study the effectiveness of ZD 1839 combined with irinotecan, leucovorin, and fluorouracil in treating patients who have locally advanced, locally recurrent, or metastatic colorectal cancer. Biological therapies such as ZD 1839 may interfere with the growth of tumor cells and slow the growth of the tumor. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining ZD 1839 with combination chemotherapy may kill more tumor cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the maximum tolerated dose of ZD 1839 in combination with irinotecan, leucovorin calcium, and fluorouracil in patients with locally advanced, locally recurrent, or metastatic colorectal cancer.

II. Determine the dose-limiting toxicity of this regimen in these patients. III. Determine the pharmacokinetics of this regimen in these patients. IV. Determine the objective response rate in patients treated with this regimen.

V. Correlate epidermal growth factor receptor expression with the probability of objective tumor response in these patients.

OUTLINE: This is a multicenter, dose-escalation study of ZD 1839.

Patients receive oral ZD 1839 daily. Beginning on day 15, patients receive irinotecan IV over 90 minutes, leucovorin calcium IV over 15 minutes, and fluorouracil IV weekly on weeks 1-2. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of ZD 1839 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, 10 additional patients are accrued to receive treatment at the MTD.

Patients are followed for 30 days.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the colon or rectum

  * Locally advanced, locally recurrent, or metastatic disease
  * Not curable by surgery and/or not amenable to radiotherapy with curative intent
  * Histological or cytological confirmation of metastatic cancer not required for patients with prior surgically resected colorectal cancer if more than 5 years elapsed between primary surgery and development of metastatic disease OR if primary cancer was stage I or II
* Prior adjuvant therapy with fluorouracil or immunotherapy for resected stage II, III, or IV disease allowed
* Measurable disease
* No known brain metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-1

Life expectancy:

* More than 12 weeks

Hematopoietic:

* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin normal
* AST/ALT no greater than 5 times upper limit of normal

Renal:

* Creatinine normal

Cardiovascular:

* No uncontrolled high blood pressure
* No unstable angina
* No symptomatic congestive heart failure
* No myocardial infarction within the past 6 months
* No serious uncontrolled cardiac arrhythmia
* No New York Heart Association class III or IV heart disease

Other:

* No active or uncontrolled infection
* No predisposing colonic or small bowel disorders with uncontrolled symptoms as indicated by more than 3 loose stools daily in patients without a colostomy or ileostomy
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or adequately treated noninvasive carcinomas
* No other concurrent medical or psychiatric condition that would preclude study
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 12 months since prior immunotherapy

Chemotherapy:

* At least 12 months since prior fluorouracil
* No prior chemotherapy for advanced colorectal cancer
* No prior irinotecan

Radiotherapy:

* No prior radiotherapy to more than 15% of bone marrow
* At least 4 weeks since prior major radiotherapy (e.g., chest or bone palliative radiotherapy)
* No concurrent radiotherapy

Surgery:

* At least 4 weeks since prior major surgery (e.g., laparotomy) and recovered
* At least 2 weeks since prior minor surgery and recovered
* No concurrent ophthalmic surgery

Other:

* No prior ZD 1839
* No other concurrent investigational or commercial agents or therapies for malignancy
* No concurrent combination antiretroviral therapy for HIV
* No concurrent oral retinoids
* No concurrent prochlorperazine on day of irinotecan administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2001-11; Primary Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles S. Fuchs, MD, Study Chair — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Result] Meyerhardt JA, Clark JW, Supko JG, Eder JP, Ogino S, Stewart CF, D'Amato F, Dancey J, Enzinger PC, Zhu AX, Ryan DP, Earle CC, Mayer RJ, Michelini A, Kinsella K, Fuchs CS. Phase I study of gefitinib, irinotecan, 5-fluorouracil and leucovorin in patients with metastatic colorectal cancer. Cancer Chemother Pharmacol. 2007 Oct;60(5):661-70. doi: 10.1007/s00280-006-0411-6. Epub 2007 Jan 11. PMID 17216531
- [Result] Wolpin BM, Clark JW, Meyerhardt JA, Earle CC, Ryan DP, Enzinger PC, Zhu AX, Blaszkowsky L, Battu S, Fuchs CS. Phase I study of gefitinib plus FOLFIRI in previously untreated patients with metastatic colorectal cancer. Clin Colorectal Cancer. 2006 Sep;6(3):208-13. doi: 10.3816/CCC.2006.n.037. PMID 17026790